CLINICAL TRIAL: NCT02433743
Title: Daily Consumption of Ready-to-use Peanut-based Therapeutic Food Increased Fat Free Mass, Improved Anemia Status But Has no Impact on Zinc Status of People Living With HIV/AIDS (PLWHA)
Brief Title: Impact of RUTF on Body Composition, Anemia and Zinc Status of PLWHA
Acronym: PLWHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cheikh Anta Diop University, Senegal (Other)
Collaborators: UNICEF (Other)
Responsible Party: Principal Investigator, Jean Louis Ndiaye, Adama Diouf, Cheikh Anta Diop University, Senegal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCheikhAntaDiop
Record Dates: First submitted 2015-04-18; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: HIV-infection/Aids; Malnutrition
Keywords: HIV/AIDS; RUTF; fat free mass; anemia; zinc; Senegal
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Malnutrition; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control group (n=33) didn't received intervention. The received the standard hospital diet
- Ready-to-use therapeutic food (RUTF) (Experimental): RUTF group (n=32) received the standard hospital diet combined with 100 g/day of RUTF
  Interventions: Dietary Supplement: Ready-to-use therapeutic food (RUTF)

INTERVENTIONS:
Dietary Supplement: Ready-to-use therapeutic food (RUTF) — HIV-infected patients were randomly allocated to receive standard hospital diet (Control: n=33), or this diet combined with 100 g/day of RUTF (RUTF: n=32). All patients was follow-up during hospitalisation and 9 week after discharge at home
  Other Names: RUTF
  Arms: Ready-to-use therapeutic food (RUTF)

SUMMARY:
A clinical trial was conducted in 65 PLWH randomly allocated to receive standard hospital diet alone (Control group: n=33), or the diet combined with 100 g/day of RUTF (RUTF group: n=32). Individual dietary intakes were measured and compared to the Recommended Dietary Allowances (RDA) for PLWH. Body composition was measured by bio-impedance analysis (BIA), hemoglobin by HemoCue and plasma zinc concentration by atomic absorption spectrometry and adjusted to infection (CRP and α1-AGP). All measures were conducted at baseline, 3 weeks and after 9 weeks home-based follow up.

DETAILED DESCRIPTION:
The sample size of the study (n=17 in each group) was calculated takin into account the mean gain of fat free mass (2.3± 2.1 kg) obtained in a study of PLWH supplemented with 43 g of RUTF/day. The randomization was performed upon admission using a computer-generated random number list (EPI INFO 6.0; Centers for Disease Control and Prevention, Atlanta).

Dietary intakes were measured during 7 consecutive days in 10 subjects of each group during the hospitalization period. Each meal served was weighed with a food scale (i-Balance 2600 Myweigh, Phoenix, USA).

Anthropometrics measurement was performed using standard procedures. Measure of height was made using height board (SECA 216, GmbH et Co, Hamburg, Germany), to the nearest millimeter. Body weight was measured with an electronic scale (SECA 877, GmbH & Co, Hamburg, Germany).

Body composition was measured using a multifrequency analyser, Xitron 4000B. The accuracy of the instrument was tested before the measurements by using a 422 ohm standard resistor purchased with the analyzer. Blood sampling was performed in the morning between 8 -10 AM into trace element-free polyethylene tubes zinc-free containing lithium heparin anticoagulant. The time of the sample collection and of the most recent food or milk intake were noted and used to adjust for this interval in the analysis of data. All the parameters were mesured in duplicate on admission, at 3 weeks and 9 weeks home based follup up.

Double entry data, and quality control of the entry were performed using Epi-Info version 3.5.1 (CDC, Atlanta, USA) and access. Statistical analysis was performed by Excel 2003 (Microsoft Corporation, Redmond, USA) and STATA / SE 11.0 (Stata Corporation, Texas, and USA). Results are expressed as mean ± standard deviation and percentage. PZ concentration was adjusted for the time interval between the last meal and the blood drawing to minimize the variability due to the known meal-related effects on PZ concentration and from infections/inflammation [28]. Zinc deficiency was defined according to IZINCG cut-off. ANOVA followed by post-hoc Bonferroni tests for pairwise comparison of means or Student's t-test were also used on dependent measures. The Pearson Chi2 test or Fisher's exact test were used to compare percentages. P values 0.05 were considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* HIV/AIDS men and women
* at any WHO stages of HIV disease,
* under ART treatment or not,
* without psychiatric illness and not diabetic

Exclusion Criteria:

* confirmed HIV-negative,
* long term physical disability
* inability to eat

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in body composition at 9 weeks | 9 weeks
  Body composition was measured using Bio-impedance analysis method at baseline, and 9 weeks home-based follow-up in both supplemented and control groups

SECONDARY OUTCOMES:
Change from baseline on anemia at 3 weeks | 3 weeks
  Hemoglobin was measured by Hemocue photometer at baseline and 3 week after admission in both supplemented and control groups
Change from baseline on anemia at 9 weeks | 9 weeks
  Hemoglobin was measured by Hemocue photometer at baseline and after 9 weeks home-based follow-up in both supplemented and control groups
Change from baseline on plasma zinc concentration at 3 weeks | 3 weeks
  Plasma zinc concentration was determined by Atomic absorption spectrometry at baseline and 3 weeks after admission in both supplemented and control groups
Change from baseline on plasma zinc concentration at 9 weeks | 9 weeks
  Plasma zinc concentration was determined by Atomic absorption spectrometry at baseline and after 9 weeks home-based follow-up in both supplemented and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Salimata Wade, Professor, Study Director — Université Cheikh Anta Diop de Dakar
Locations (1):
- University Cheikh Anta Diop, Dakar, Senegal

REFERENCES:
- [Derived] Diouf A, Badiane A, Manga NM, Idohou-Dossou N, Sow PS, Wade S. Daily consumption of ready-to-use peanut-based therapeutic food increased fat free mass, improved anemic status but has no impact on the zinc status of people living with HIV/AIDS: a randomized controlled trial. BMC Public Health. 2016 Jan 4;16:1. doi: 10.1186/s12889-015-2639-8. PMID 26728978